CLINICAL TRIAL: NCT04592042
Title: Intervention to Improve Coping With Negative Emotions in Patients With Psychotic Disorders: Feasibility and Efficacy of an Emotion-oriented Cognitive-behavioural Group Intervention ("Feel-Good-Group").
Brief Title: Intervention to Improve Coping With Negative Emotions in Patients With Psychosis (Feel-Good-Study)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Prof. Dr. Andreas Bechdolf (Chair of hospital), Vivantes Hospital Am Urban Berlin (Unknown); Prof. Dr. Nikola Stenzel (Collaboration partner), Berlin Psychological University, Berlin (Unknown); Dr. Karolina Leopold (Senior physician), Vivantes Hospital Am Urban Berlin (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Stephanie Mehl, Principal Investigator, Managing Psychologist, Philipps University Marburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Feel-Good-Study
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Early Psychosis; Delusions; Emotional Distress; Self Esteem
Keywords: Psychosis; Cognitive behavioral therapy; Group therapy; targeted therapy; emotion regulation; emotional stability
MeSH Terms: conditions — Psychotic Disorders; Delusions; Emotional Regulation | interventions — Inosine Monophosphate

STUDY DESIGN:
Intervention Model Description: A single group of patients will be enrolled in the study.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feel-Good-Group (Experimental): Pre-post assessment of feasibility and putative efficacy of an emotion-oriented cognitive-behavioral group intervention over 8 sessions and four weeks.
  Interventions: Behavioral: Feel-Good- Group

INTERVENTIONS:
Behavioral: Feel-Good- Group — Eight sessions of group intervention focussing on information on emotion regulation, training of emotion regulation techniques and mindfulness.
  Other Names: Emotion-oriented version of Cognitive Behavior Therapy for psychosis in group format for inpatients with psychosis

SUMMARY:
The aim of the present single-centered pre-post study is to assess the feasibility and to investigate the putative efficacy of an emotion-oriented group intervention for patients with psychosis. Patients with early psychosis in an inpatient unit receive a manualized group intervention focussing on emotional stability and emotion regulation (8 weekly sessions). Assessment will be performed at pre-therapy, post-therapy (after eight sessions and four weeks) and after a follow-up period of 12 weeks (8 weeks post therapy) and includes personal therapy goals and their realization, psychopathology, social functioning and emotion regulation skills as a putative mediator of change.

DETAILED DESCRIPTION:
The aim of the present single-centered pre-post study is to assess the feasibility and to investigate the putative efficacy of an emotion-oriented cognitive-behavioral group intervention for patients with psychosis.

Patients with psychosis in an inpatient unit are informed on the study and written consent is obtained. At start of therapy, psychopathological interviews and self-report questionnaires are performed. Participants are reassessed after the intervention of 8 sessions (approximately 8 weeks) and after a follow-up period of 8 additional weeks).

Patients are enrolled in a manualized group therapy over 8 sessions including 7 modules. In the first session, group rules are obtained and individual therapy goals are elaborated and developed for each patient. In the next seven sessions, in each session a new module is presented to the patient and the skills are trained in training sessions and role plays.

Module 1 informs on emotions and their role in mental health, module 2 informs on techniques/skills in order to cope with negative emotions more generally. In module 3, mindfulness is presented as a technique to reduce the impact of negative emotions on the patients' life and practised. In module 4, patients learn skills on how to reduce their vulnerability for negative emotions in general. In Module 5, patients learn skills on how to cope with anger, Module 6 teaches skills on how to cope with guilt and shame, Module 7 is presented in the last session and includes skills on how to improve general emotional stability and to prevent relapse.

Training: Therapists are psychologists or psychiatrists that are currently in postgraduate training of Cognitive Behavior Therapy and received 8 sessions of additional training by the study PI.

Primary outcome variables are attainment of the individual therapy goals of the patient (Goal Attainment Scale) and reduced general psychopathology (PANSS total score) after 8 sessions therapy. Secondary outcomes are depressive symptoms (Calgary Depression Scale for Schizophrenia), social functioning (Role functioning scale), self-reported delusions (Peters et al. delusions inventory), self-reported persecutory delusions (Paranoia checklist), emotion regulation skills (Emotion Regulation Skills Questionnaire, Emotion regulation questionnaire, Emotion Regulation Inventory), self-esteem (Rosenberg Self-esteem Questionnaire) and the Beliefs About Stress Scale (BASS). Furthermore, patients are asked to assess feasibility and acceptance of the group intervention. Emotion regulation skills and self-esteem are also tested as putative mediators of change.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, psychotic disorder, bipolar disorder with psychotic symptoms using the International Classification of Diseases-10 (ICD-10 (Codes: F 20.x, F21.x, F22.x, F 23.x, F 25, F30.x, F 31.x ) verified by the Structured Clinical Interview for Diagnostic and Statistical Manual for Mental Disorders 5-Clinical Version (SCID-5-CV) Beesdo-Baum et al., 2019) transformed to ICD-10.
* first psychotic episode in the last five years
* written informed consent provided by patient or legal guardian
* estimated verbal intelligence of at least 80 IQ-scores estimated with the German Mehrfachwahlwortschatztest (MWT-B, Lehrl et al., 2005)

Exclusion Criteria:

* acute suicidality
* diagnosis of dementia (verified by the SCID-5-CV interview and patient documentation)

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Goal attainment scale (GAS, Kiresuk & Sherman, 1968) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Patients select in an individual session with their therapist their most important therapy goal and mark on a scale from 0-100, whether it is reached at the present day. The mean score will be used (range between 0 and 100 with higher scores indicating higher values)
Positive and Negative Scale Total score (Kay et al., 1992) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Interview to assess positive symptoms, negative symptoms and general psychopathology in the last week. Range 30-210 with higher scores indicating more pronounced distress.

SECONDARY OUTCOMES:
Psychotic Symptoms Rating Scale delusions subscale (PSYRATS, Haddock et al., 1999) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Interview to assess present delusions and hallucinations, the related distress, conviction rate, frequency and problems in daily life caused by the symptoms. Range 0 - 28 with higher scores indicating more pronounced delusions
Calgary Depression Scale for Schizophrenia (CDSS; Mueller et al., 1999) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Interview to assess depressive symptoms. Range between 0 and 44 with higher scores indicating more pronounced depressive symptoms.
Peters et al, Delusions Inventory (PDI; Lincoln, Keller & Rief, 2009) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-report questionnaire assessing endorsement of 21 delusions, frequency, distress and conviction rate in the last week. Grand total score, range between 0 and 312 with higher scores indicating more pronounced self-rated delusions.
Role Functioning Scale (RFS; Goodman et al., 1999) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Interview to assess role functioning, number of close relationship, community integration, work integration and community integration. Mean score of all four scores: range between 0 and 12 with higher scores indicating more pronounced functioning.
Paranoia checklist (Freeman et al., 2005) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-report assessment of persecutory delusions, frequency, distress and conviction. The total score will be used, range between 0 and 270 with higher scores indicating more pronounced paranoid symptoms.
Emotion Regulation Skills Questionnaire (ERSQ; Berking & Znoj, 2008) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-reported assessment of emotion regulation skills (e.g. mindfulness, suppression), Total score: range between 0 and 108 with higher scores indicating more elaborated emotion regulation skills.
Emotion Regulation Questionnaire (ERQ; Gross & John, 2003) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-reported assessment of emotion regulation skills (e.g. cognitive restructuring). The total score will be used (range 10-70) with higher scores indicating more pronounced emotion regulation skills.
Emotion Regulation Inventory (ERI; Koenig, 2011) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-reported assessment of emotion regulation skills (e.g. distraction). The total score will be used (range between 10 and 70 with higher scores indicating more pronounced emotion regulation skills.
Rosenberg Self-Esteem Scale (RSE; Collani & Herzberg, 2003) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-reported assessment of global self-worth and self-esteem. The total score will be used (range between 0-30) with higher scores indicating good self-esteem.
Beliefs About Stress Scale (BASS; Laferton et al., 2016) | Change between start of therapy and end of therapy (approximately 8 weeks).
  Self-reported assessment of illness perception. The negative stress beliefs score will be used (range between 0 and 32) with higher scores indicating more pronounced negative beliefs about stress.
Feasibility and acceptance of therapy (Lincoln et al., 2012) | Change between start of therapy and end of therapy(approximately 8 weeks).
  Self-reported assessment of feasibility and acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nikola M Stenzel, Ph. D., Study Chair — Psychologische Hochschule Berlin; Andreas Bechdolf, MD, Study Director — Vivantes Klinikum Am Urban, Berlin; Karolina Leopold, MD, Study Chair — Vivantes Klinikum Am Urban, Berlin
Locations (1):
- University of Marburg, Faculty of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized data of the study on an online repository (Open Science Foundation)
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available 6 month after the end of the study (September 2023)
Access Criteria: no criteria
URL: http://www.osf.io

REFERENCES:
- [Derived] von Hardenberg L, Leopold K, Pfennig A, Kuhn C, Kallenbach M, Aliakbari N, Mehl S, Bechdolf A. Subjective experiences of an acceptance and mindfulness-based group intervention (Feel-Good-Group) in young people with early psychosis. Front Psychiatry. 2024 Oct 7;15:1369629. doi: 10.3389/fpsyt.2024.1369629. eCollection 2024. PMID 39435124
- [Derived] von Hardenberg L, Leopold K, Stenzel N, Kallenbach M, Aliakbari N, Bechdolf A, Mehl S. Feasibility and efficacy of an acceptance and mindfulness-based group intervention for young people with early psychosis (Feel-Good group). Front Psychiatry. 2022 Sep 16;13:943488. doi: 10.3389/fpsyt.2022.943488. eCollection 2022. PMID 36186856